CLINICAL TRIAL: NCT05554367
Title: Palbociclib and Binimetinib in RAS-Mutant Cancers: A ComboMATCH Treatment Trial
Brief Title: Palbociclib and Binimetinib in RAS-Mutant Cancers, A ComboMATCH Treatment Trial
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2022-07266; NCI-2022-07266 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EAY191-A3 (Other: Alliance for Clinical Trials in Oncology); EAY191-A3 (Other: CTEP); U10CA180821 (NIH)
Record Dates: First submitted 2022-09-22; First posted 2022-09-26 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-09

CONDITIONS: Exocrine Pancreas Carcinoma; Malignant Solid Neoplasm; Ovarian Low Grade Serous Adenocarcinoma; Stage IV Ovarian Cancer AJCC v8; Stage IV Pancreatic Cancer AJCC v8
MeSH Terms: conditions — Pancreatic Neoplasms; Ovarian Neoplasms | interventions — binimetinib; Biopsy; Specimen Handling; Magnetic Resonance Spectroscopy; palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Combination Cohorts 1, 2, 3, 4 (palbociclib, binimetinib) (Experimental): Patients receive palbociclib PO QD on days 1-21 and binimetinib PO BID on days 1-28 of each cycle. throughout the trial. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity for up to 3 years. Patients may also undergo biopsy at screening and undergo MRI, CT, bone scan, and collection of blood samples during screening, on study, and/or during follow up.
  Interventions: Drug: Binimetinib; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Drug: Palbociclib
- Monotherapy Cohort 1 (binimetinib) (Experimental): Patients receive binimetinib PO BID daily, in the absence of disease progression or unacceptable toxicity, for up to 3 years. Patients who experience disease progression may elect to migrate to the combination cohort. Patients may also undergo biopsy at screening and undergo MRI, CT, bone scan, and collection of blood samples during screening, on study, and/or during follow up.
  Interventions: Drug: Binimetinib; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Drug: Binimetinib — Given PO
  Other Names: ARRY 162; ARRY 438162; ARRY-162; ARRY-438162; ARRY162; ARRY438162; MEK 162; MEK-162; MEK162; Mektovi
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Scan — Undergo bone scan
  Other Names: Bone Scintigraphy
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Palbociclib — Given PO
  Other Names: 6-Acetyl-8-cyclopentyl-5-methyl-2-((5-(piperazin-1-yl)pyridin-2-yl)amino)-8h-pyrido(2,3-d)pyrimidin-7-one; Ibrance; PD 0332991; PD 332991; PD 991; PD-0332991; PD0332991
  Arms: Combination Cohorts 1, 2, 3, 4 (palbociclib, binimetinib)

SUMMARY:
This phase II ComboMATCH treatment trial evaluates the effectiveness of palbociclib and binimetinib in treating patients with RAS-mutated cancers. Palbociclib and binimetinib are both in a class of medications called kinase inhibitors. They work by blocking the action of abnormal proteins that signals cancer cells to multiply. This trial may help researchers understand if giving the combination of palbociclib and binimetinib can help improve the amount of time before the cancer grows in patients with patients with low grade serous ovarian cancer who have certain changes in the tumor DNA. This trial may also help researchers understand if giving the combination of palbociclib and binimetinib can help improve outcomes among patients with low grade serous ovarian cancer who have previously received a MEK inhibitor. For patients with other tumors, with the exception of lung cancer, colon cancer, melanoma and low grade serous ovarian cancers, this trial may help researchers understand if giving the combination of palbociclib and binimetinib can improve the clinical outcome of survival without progression in patients who have certain changes in their tumor's DNA.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether palbociclib and binimetinib combination therapy improves progression free survival (PFS) compared to binimetinib alone in patients with MEK-inhibitor naive low-grade serous ovarian cancer (LGSOC) harboring MAP kinase activation (KRAS/NRAS/non BRAF V600E mutation). (Cohort 1) II. To determine whether palbociclib and binimetinib improves clinical activity in comparison to historical control, as measured by objective response rate (ORR), in women with LGSOC whose disease has previously progressed on a MEK inhibitor. (Cohort 2) III. To determine whether palbociclib and binimetinib combination therapy improves the objective response rate compared to historical control in patients with pancreatic cancer harboring any KRAS/NRAS/HRAS mutation or non-BRAF V600E aMOIs or rare RAF fusion. (Cohort 3) IV. To determine whether palbociclib and binimetinib combination therapy improves objective response rate compared to historical control in patients with tumors harboring any KRAS/NRAS/HRAS mutations or non-BRAF V600E aMOIs or rare RAF fusions (excluding LGSOC, non-small cell lung cancer [NSCLC], colorectal cancer, pancreatic cancer and melanoma). (Cohort 4)

SECONDARY OBJECTIVES:

I. To determine whether palbociclib and binimetinib combination therapy improves objective response rate (ORR), overall survival (OS), duration of response (DOR), and disease control rate (DCR) compared to binimetinib alone in patients with MEK inhibitor-naïve LGSOC. (Cohort 1) II. Conduct whole-exome sequencing to evaluate concordance with the designated laboratory result. (Cohort 1) III. To assess the clinical activity of palbociclib and binimetinib as measured by PFS, OS, DOR, and DCR in women with LGSOC whose disease has previously progressed on a MEK inhibitor. (Cohort 2) IV. Conduct whole-exome sequencing to evaluate concordance with the designated laboratory result. (Cohort 2) V. To assess the clinical activity of palbociclib and binimetinib as measured by PFS, OS, DOR, and DCR in patients with RAS mutated pancreatic cancer. (Cohort 3) VI. Conduct whole-exome sequencing to evaluate concordance with the designated laboratory result. (Cohort 3) VII. To assess the clinical activity of palbociclib and binimetinib as measured by PFS, OS, DOR, and DCR in patients with RAS mutated cancers, excluding LGSOC, NSCLC, colorectal cancer (CRC), pancreatic cancer and melanoma. (Cohort 4) VIII. Conduct whole-exome sequencing to evaluate concordance with the designated laboratory result. (Cohort 4)

EXPLORATORY OBJECTIVES:

I. Explore thymidine kinase 1 (TK1) activity in response to palbociclib. (Cohort 1) II. Assess the correlation between presence of KRAS mutation and activity of both monotherapy and the combination. (Cohort 1) III. Conduct ribonucleic acid (RNA)-sequencing (seq) to assess determinants of response and resistance. (Cohort 1) IV. Explore changes in plasma RAS allelic burden in KRAS-mutated tumors using circulating tumor deoxyribonucleic acid (ctDNA) and correlate changes with clinical activity. (Cohort 1) V. Explore TK1 activity in response to palbociclib.(Cohort 2) VI. Assess the correlation between presence of KRAS mutation and activity of the combination. (Cohort 2) VII. Conduct RNA-seq to assess determinants of response and resistance. (Cohort 2) VIII. Explore changes in plasma RAS allelic burden in KRAS-mutated tumors using ctDNA and correlate changes with clinical activity. (Cohort 2) IX. Explore TK1 activity in response to palbociclib. (Cohort 3) X. Evaluate changes in deoxyribonucleic acid (DNA), RNA and ctDNA to evaluate concordance with the designated laboratory result and to assess determinants of response, signatures of intrinsic resistance or response and the plasma RAS allelic burden in relation to treatment response, respectively. (Cohort 3) XI. Explore TK1 activity in response to palbociclib. (Cohort 4) XII. Evaluate changes in DNA, RNA and ctDNA to evaluate concordance with the designated laboratory result and to assess determinants of response, signatures of intrinsic resistance or response and the plasma RAS allelic burden in relation to treatment response, respectively. (Cohort 4)

OUTLINE: Patients with KRAS, NRAS, non-BRAF V600E aMOIs or rare RAF fusions LGSOC, naïve to MEK or CDK4/6 inhibitor therapy are randomized to either combination cohort 1 or monotherapy cohort 1. Patients with LGSOC who have received prior MEK inhibitor therapy are assigned to combination cohort 2. Patients with KRAS/NRAS/HRAS/non-V600E a MOIs or rare RAF fusion pancreatic cancer are assigned to combination cohort 3. Patients with all other KRAS/NRAS/HRAS, non -BRAF V600E a MOIs or rare FAR fusion tumor types (excluding LGSOC, NSCLC, CRC, pancreatic, and melanoma) are assigned to combination cohort 4.

COMBINATION COHORTS 1, 2, 3, 4: Patients receive palbociclib orally (PO), once per day (QD) on days 1-21 and binimetinib PO twice per day (BID) on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity for up to 3 years. Patients may also undergo biopsy at screening and undergo magnetic resonance imaging (MRI), computed tomography (CT), bone scan, and collection of blood samples during screening, on study, and/or during follow up.

MONOTHERAPY COHORT 1: Patients receive binimetinib PO BID daily, in the absence of disease progression or unacceptable toxicity, for up to 3 years. Patients who experience disease progression may elect to migrate to the combination cohort. Patients may also undergo biopsy at screening and undergo MRI, CT, bone scan, and collection of blood samples during screening, on study, and/or during follow up.

After completion of study treatment, patients are followed up every 3 months for up to 3 years following registration.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have enrolled onto EAY191 and must have been given a treatment assignment to ComboMATCH to EAY191-A3 based on the presence of an actionable mutation as defined in EAY191.
* GENERAL ComboMATCH EAY191 REGISTRATION INCLUSION CRITERIA:
* Patients must be enrolled on the EAY191 registration study and be assigned to this protocol by EAY191
* Patients must have KRAS/NRAS/HRAS or RAF mutations or rare RAF fusions as determined by the ComboMATCH screening assessment
* Patients with low grade serous ovarian cancer who have progressed on a prior MEK inhibitor are not required to have a KRAS/NRAS/HRAS or BRAF alteration
* Patients must not have a BRAF V600E alteration as determined by the ComboMATCH screening assessment
* Patients with a tumor harboring KRAS G12C mutation will be eligible either after they have received a G12C inhibitor or can be enrolled if they do not meet eligibility for a G12C inhibitor. However, patients with tumors harboring KRAS G12C mutation will be prioritized for a G12C inhibitor-based substudy if eligible
* Patients must have disease that can be safely biopsied and agree to a pre-treatment biopsy or have archival tissue available from within 12 months prior to registration
* Please note the current actionable marker of interest (aMOI)/actionable alteration list for this treatment trial can be found on the Cancer Trials Support Unit (CTSU) website
* EAY191-A3 IELIGIBILITY CRITERIA:
* Histologically confirmed cancer for each cohort for which curable treatment modalities are not an option. Rare BRAF fusions and non-BRAF V600E aMOIs are acceptable. RB1 mutations or two copy RB1 deletions are excluded
* Tumor tissue must be available:

  * Adequate archival tumor specimen (obtained within 12 months of EAY191 registration which has not had a Response Evaluation Criteria in Solid Tumors (RECIST) response, complete response (CR) or partial response (PR), to any intervening therapy after collection of the tissue) must be available with formalin-fixed paraffin-embedded tumor tissue (blocks or slides) OR
  * Consent to a new tumor tissue biopsy which is not a representative target lesion. This lesion must be amenable to a minimal risk image-guided or direct vision biopsy A new biopsy is preferred but is not required for enrollment in EAY191-A3 if sufficient archival tissue is available as described above
* Measurable disease per RECIST 1.1. Of note, in the case when a baseline biopsy is done after scans are obtained, a lesion separate from one that is biopsied needs to be measurable per RECIST 1.1. All radiologic studies must be performed within 28 days prior to registration
* COHORT 1: Low grade serous ovarian cancer with KRAS, NRAS non-BRAF V600E aMOIs or rare RAF fusions are acceptable
* COHORT 1: No prior MEK inhibitor or CDK4/6 inhibitor therapy
* COHORT 1: Any number of prior therapies permitted
* COHORT 1: No major surgery within 4 weeks (excluding placement of vascular access), minor surgery within 2 weeks, or palliative radiotherapy within 2 weeks prior to registration
* COHORT 1: No prior cancer-directed therapy within 28 days prior to registration. Patients may have received cancer-directed hormonal therapy up to 14 days prior to registration
* COHORT 2: Low grade serous ovarian cancer
* COHORT 2: Prior progression of disease on a MEK inhibitor (prior binimetinib permitted)
* COHORT 2: If patient has previously received binimetinib, they cannot have required dose reduction or discontinuation of binimetinib due to adverse events
* COHORT 2: No prior receipt of a CDK4/6 inhibitor
* COHORT 2: No major surgery within 4 weeks (excluding placement of vascular access), minor surgery within 2 weeks, or palliative radiotherapy within 2 weeks prior to registration
* COHORT 2: No prior cancer-directed therapy within 28 days prior to registration. Patients may have received cancer-directed hormonal therapy up to 14 days prior to registration
* COHORT 3: Pancreatic cancer with KRAS/NRAS/HRAS, non-BRAF V600E aMOIs or rare RAF fusions are acceptable
* COHORT 3: No prior MEK inhibitor (MEKi) and CDK4/6i therapy
* COHORT 3: Progression after at least one line of prior therapy as long as there is no standard therapy available or acceptable to patients that is thought to be of benefit
* COHORT 3: Any number of prior therapies are permitted
* COHORT 3: No major surgery within 4 weeks (excluding placement of vascular access), minor surgery within 2 weeks, or palliative radiotherapy within 2 weeks prior to registration
* COHORT 3: No prior cancer-directed therapy within 28 days prior to registration. Patients may have received cancer-directed hormonal therapy up to 14 days prior to registration
* COHORT 4: KRAS/NRAS/HRAS non-BRAF V600E aMOIs or rare RAF fusions are acceptable
* COHORT 4: No prior MEKi and CDK4/6i therapy and progression after at least one line of prior therapy, as long as there is no standard therapy available or acceptable to patients that is thought to be of benefit
* COHORT 4: Any number of prior therapies are permitted
* COHORT 4: No more than 6 patients with a given tumor type allowed in this cohort
* COHORT 4: Any tumor type, except: LGSOC/NSCLC/CRC/pancreatic/melanoma
* COHORT 4: No major surgery within 4 weeks (excluding placement of vascular access), minor surgery within 2 weeks, or palliative radiotherapy within 2 weeks prior to registration
* COHORT 4: No prior cancer-directed therapy within 28 days prior to registration. Patients may have received cancer-directed hormonal therapy up to 14 days prior to registration
* Not pregnant and not nursing, because this study involves investigational agents whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown. Therefore, for women of childbearing potential only, a negative pregnancy test done =< 7 days prior to registration is required
* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status < 2
* Absolute neutrophil count (ANC) >= 1,500/mm^3
* Platelet count >= 100,000/mm^3
* Hemoglobin > 9 g/dL
* Creatinine =< 1.5 x upper limit of normal (ULN) or calculated (calc.) creatinine clearance >= 30 mL/min as calculated by the Cockcroft-Gault formula
* Total bilirubin =< 1.5 x upper limit of normal (ULN). Patients with Gilbert syndrome may enroll if total bilirubin (bili) < 3 mg/dL (51 micromole/L)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 2.5 x upper limit of normal (ULN)
* Creatine phosphokinase (CPK) =< 2.5 x ULN
* Patients must be able to swallow oral formulations of the agents
* No history of interstitial lung disease. No history of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan
* Patients should not have history of bowel perforation or intestinal fistulas in the last 6 months
* No patients with the inability to swallow oral medications or impaired gastrointestinal absorption due to gastrectomy or active inflammatory bowel disease
* No active skin disorder that has required systemic therapy within the past 1 year
* No history of rhabdomyolysis
* No concurrent ocular disorders including:

  * Subjects with history of glaucoma, history of retinal vein occlusion (RVO), predisposing factors for RVO, including uncontrolled hypertension, uncontrolled diabetes
  * Subject with history of retinal pathology or evidence of visible retinal pathology that is considered a risk factor for RVO, intraocular pressure > 21 mm Hg as measured by tonometry, or other significant ocular pathology, such as anatomical abnormalities that increase the risk for RVO
  * Subjects with a history of corneal erosion (instability of corneal epithelium), corneal degeneration, active or recurrent keratitis, and other forms of serious ocular surface inflammatory conditions
* No patients with a history of hypersensitivity to any of the study drug(s)
* No prior allogeneic stem cell or solid organ transplantation
* Central nervous system (CNS) metastases must have been treated with local therapy (surgery, radiation, ablation) and patient off of systemic steroids, and brain metastases stable for at least 1 month
* No residual Common Terminology Criteria for Adverse Events (CTCAE) >= grade 2 toxicity from any prior anticancer therapy, with the exception of grade 2 alopecia
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients whose left ventricular ejection fraction (LVEF) has been evaluated by echocardiography (ECHO)/multigated acquisition scan (MUGA) are excluded if the most recent exam shows an LVEF < 50%
* Chronic concomitant treatment with strong inhibitors of CYP3A4 is not allowed on this study. Patients on strong CYP3A4 inhibitors must discontinue the drug for 14 days prior to registration on the study
* Chronic concomitant treatment with strong CYP3A4 inducers is not allowed. Patients must discontinue the drug 14 days prior to the start of study treatment
* No exposure to P-glycoprotein (P-gp) inhibitors or inducers within 14 days prior to the first dose and during the course of therapy
* Patients treated with Cohort 1 control treatment binimetinib who experience disease progression may elect to migrate to cohort 2 and receive combination treatment with palbociclib and binimetinib. Patients who choose to do so must meet laboratory values and performance status requirements as above and must be begin treatment within 21 days. For patients who migrate from cohort 1 to cohort 2, the 28-day window restricting prior anti-cancer directed therapies does not apply to prior binimetinib. A new biopsy will not be required for migration, but the optional biopsy at disease progression should be encouraged

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Estimated)
Dates: Start 2023-12-13 (Actual); Primary Completion 2026-08-26 (Estimated); Study Completion 2026-08-26 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) (Cohort 1) | Time from randomization date until the time of disease progression or death due to any cause, assessed at 6, 12, 18, 24, and 30 months
  Will compare the PFS distributions between those treated with palbociclib and binimetinib vs. binimetinib alone. PFS will be compared between the two treatment arms using Kaplan-Meier methods. The hazard ratio, median PFS, and estimated PFS rates at 6, 12, 18, 24, and 30 months will be estimated along with corresponding 95% confidence intervals. A log-rank test will be used to compare the PFS distributions between the two treatment arms in this cohort. In an ancillary manner, Cox proportional hazards models will also be used to assess the impact of treatment arm on PFS when stratifying on the stratification factors.
Objective response rate (ORR) (Cohort 2) | Up to 3 years
  The Simon optimal design used to evaluate efficacy in terms of the objective response rate after treatment in this population will use a two-stage design.
ORR (Cohort 3) | Up to 3 years
  The Simon minimax design used to evaluate efficacy in terms of the objective response rate after treatment in this population will use a two-stage design.
ORR (Cohort 4) | Up to 3 years
  The Simon minimax design used to evaluate efficacy in terms of the objective response rate after treatment in this histology/tumor agnostic population will use a two-stage design.

SECONDARY OUTCOMES:
Objective response (Cohort 1) | Up to 3 years
  Objective response by Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1 criteria will be estimated using ORR where ORR is defined as the number of evaluable patients achieving a response (partial response [PR] or complete response [CR] per RECIST v1.1) during treatment with study therapy divided by the total number of evaluable patients. Rates of response will be compared between treatment arms using a chi-square test (or Fisher's exact test as needed). Point estimates will be generated for objective response rates within each arm along with 95% confidence intervals using the Clopper-Pearson method.
PFS (Cohorts 2, 3, 4) | From study entry to the first of either disease progression or death from any cause, assessed up to 3 years
  Disease progression will be determined based on RECIST 1.1 criteria. PFS will be estimated using the Kaplan-Meier method. The median PFS and corresponding 95% confidence interval will be reported. Patients will be censored at the last disease assessment date if they were alive and progression-free at the time of their last assessment.
Overall survival (OS) (All Cohorts) | From registration until death due to any cause, assessed up to 3 years
  Patients who are alive at last follow-up will be censored at that time point. The distribution of OS will be estimated using method of Kaplan-Meier. The median OS and 95% confidence interval will be reported.
Duration of response (DoR) (All Cohorts) | From patient's earliest best objective status to earliest date of progression, assessed up to 3 years
  DoR is defined for all evaluable patients who have achieved an objective response as time from the patient's earliest best objective status is first noted as either a CR or PR to the earliest date progression is documented, or death if no prior evidence of disease progression. The distribution of DoR will be estimated using the method of Kaplan-Meier.
Disease control (All Cohorts) | Up to 3 years
  Disease control will be estimated using disease control rate (DCR), which is defined as the patients who experience CR or PR per RECIST 1.1 or maintain stable disease for at least 6 months after randomization divided by the total number of evaluable patients. DCR will be evaluated within cohorts, and for cohort 1 this will also be compared between treatment arms using a chi square test. Point estimates will be generated for disease control rates within each arm along with 95% confidence intervals using the Clopper-Pearson method.
Incidence of adverse events (AE) (All Cohorts) | Up to 3 years
  All eligible patients that have initiated treatment will be considered evaluable for assessing AE rate(s). Patients will be evaluated for adverse events using the National Cancer Institute's Common Toxicity Criteria for Adverse Events version 5.0. The maximum grade for each type of AE will be recorded for each patient, and frequency tables will be reviewed to determine patterns. Additionally, the relationship of the AE(s) to the study treatment will be taken into consideration.

OTHER OUTCOMES:
TK1 activity (Cohorts 1 and 2) | Up to 3 years
  Will explore TK1 activity before vs. after treatment and how this corresponds and correlates to clinical outcomes after treatment with palbociclib.
KRAS mutations (Cohorts 1 and 2) | Up to 3 years
  Will characterize patients based on presence of KRAS mutations and how these correspond to efficacy outcomes such as PFS and response to treatment. Further, for cohort 1, will also evaluate how presence of this mutation influences outcomes in patients treated with monotherapy vs. the combination therapy. If numbers are sufficient, will also explore if KRAS mutation has any role as an effect modifier in this setting.
Determinants of response and resistance (Cohorts 1 and 2) | Up to 3 years
  Will conduct whole-exome sequencing and ribonucleic acid (RNA)-sequencing at baseline, and on optional biopsy upon progression to assess determinants of response and resistance. For cohort 1, concordance of diagnostic tumor mutation profile generated by the designated laboratory, the pre-treatment biopsy mutation profile, and the pre-treatment circulating tumor deoxyribonucleic acid (ctDNA) mutation profile will be assessed.
Changes in plasma RAS allelic burden in KRAS-mutated tumors (Cohorts 1 and 2) | Up to 3 years
  Will explore changes in plasma RAS allelic burden in KRAS-mutated tumors using ctDNA and correlate changes with clinical activity.
TK1 activity (Cohorts 3 and 4) | Up to 3 years
  Will explore TK1 activity before vs. after treatment and how this corresponds and correlates to clinical outcomes after treatment with palbociclib.
Determinants of response (Cohorts 3 and4) | Up to 3 years
  Will evaluate change in deoxyribonucleic acid (DNA), RNA, and ctDNA. Concordance of diagnostic tumor mutation profile generated by the designated laboratory, the pre-treatment biopsy mutation profile, and the pre-treatment ctDNA mutation profile will be assessed.
Signatures of intrinsic resistance or response (Cohorts 3 and 4) | Up to 3 years
  Will evaluate change in DNA, RNA, and ctDNA. Concordance of diagnostic tumor mutation profile generated by the designated laboratory, the pre-treatment biopsy mutation profile, and the pre-treatment ctDNA mutation profile will be assessed.
Plasma RAS allelic burden in in relation to response (Cohorts 3 and 4) | Up to 3 years
  Will evaluate change in DNA, RNA, and ctDNA. Concordance of diagnostic tumor mutation profile generated by the designated laboratory, the pre-treatment biopsy mutation profile, and the pre-treatment ctDNA mutation profile will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey I Shapiro, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (267):
- United States (266):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - UC San Diego Health System - Encinitas, Encinitas, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - UC San Diego Medical Center - Hillcrest, San Diego, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Cancer Care and Hematology-Fort Collins, Fort Collins, Colorado
  - UCHealth Greeley Hospital, Greeley, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - UM Sylvester Comprehensive Cancer Center at Aventura, Aventura, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Advocate Good Shepherd Hospital, Barrington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - AMG Crystal Lake - Oncology, Crystal Lake, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Northwestern Medicine Glenview Outpatient Center, Glenview, Illinois
  - Northwestern Medicine Grayslake Outpatient Center, Grayslake, Illinois
  - Advocate South Suburban Hospital, Hazel Crest, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Condell Memorial Hospital, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Advocate Outpatient Center - Oak Lawn, Oak Lawn, Illinois
  - Northwestern Medicine Orland Park, Orland Park, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Advocate High Tech Medical Park, Palos Heights, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Mercyhealth Cancer Institute - Rockford, Rockford, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Waukee Clinic, Waukee, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - MaineHealth Maine Medical Center- Scarborough, Scarborough, Maine
  - MaineHealth Cancer Care and IV Therapy - South Portland, South Portland, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - UPMC Western Maryland, Cumberland, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - OSF Saint Francis Hospital and Medical Group, Escanaba, Michigan
  - Corewell Health Farmington Hills Hospital, Farmington Hills, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo Cancer Center, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Michigan Healthcare Professionals Pontiac, Pontiac, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Mount Sinai Hospital, New York, New York
  - Upstate Cancer Center at Oswego, Oswego, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Upstate Cancer Center at Verona, Verona, New York
  - Duke University Medical Center, Durham, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Miami Valley Hospital South, Centerville, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Premier Blood and Cancer Center, Dayton, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Columbus Oncology and Hematology Associates, Dublin, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Miami Valley Cancer Care and Infusion, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - UPMC Altoona, Altoona, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - UPMC Hillman Cancer Center at Rocco And Nancy Ortenzio Cancer Pavilion, Mechanicsburg, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - UPMC Hillman Cancer Center - Monroeville, Monroeville, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Hendrick Medical Center, Abilene, Texas
  - Houston Methodist Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Methodist Willowbrook Hospital, Houston, Texas
  - Houston Methodist West Hospital, Houston, Texas
  - Houston Methodist Saint John Hospital, Nassau Bay, Texas
  - Houston Methodist Sugar Land Hospital, Sugar Land, Texas
  - Houston Methodist The Woodlands Hospital, The Woodlands, Texas
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Aurora Saint Luke's South Shore, Cudahy, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Mercyhealth Hospital and Cancer Center - Janesville, Janesville, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Eastpark Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
- Centro Comprensivo de Cancer de UPR, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm